CLINICAL TRIAL: NCT00352456
Title: Psychobiological Mechanisms of Behavioral Dysregulation
Brief Title: Psychological Mechanisms of Behavioral Dysregulation
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040271; 04-M-0271
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Neural Systems; Psychopathology
Keywords: Amygdala; Facial Affect; Instrumental Learning; Psychopathy; Emotion; Orbitofrontal Cortex; Healthy Volunteer; HV
MeSH Terms: conditions — Antisocial Personality Disorder

SUMMARY:
This study is directed toward a better understanding of how the brain regulates emotions and social and antisocial behavior. It will look at the use of the orbital frontal cortex and amygdala of the brain. Brain changes are involved in solving conflicts and the feelings that such conflicts produce. Conflicts may occur with other people or with general social rules. The researchers' expectations are that the findings will be useful in developing therapies that may improve people's ability to solve social conflicts and reduce antisocial behavior.

Adults ages 20 to 50 years of age with psychopathy and a second set of comparison adults, all of whom have been released from the Fairfax County Adult Detention Center, may be eligible for this study.

The neurocognitive component of the study, the one pertaining to performance of various tasks, will involve 20 adults with psychopathy and 20 comparison adults. The neuroimaging component, in which a magnetic resonance imaging (MRI) scan is used, will involve 18 adults and 18 comparison adults. Two visits by participants will be entailed. At the first visit, patients will undergo the following procedures and tests:

* Physical examination
* Test of vital signs, lying and standing.
* Electrocardiogram.
* Collection of blood for chemistry and hematology.
* Urinalysis and liver function tests.
* Screen for HIV and hepatitis.
* Pregnancy test, if applicable, at the first visit and at all further visits.

Depending on the group to which they are assigned, at the second visit, patients will undergo an MRI scan or take part in a variety of computer-based tasks to measure different forms of thinking skills, emotional responses, and decision making. During the MRI scan, patients will lie still on a table that will slide into the enclosed tunnel of the MRI scanner. They will be asked to lie as still as possible. As the scanner takes pictures, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. Patients will be able to communicate with the MRI staff at all times during the scan, and they may ask to be moved out of the machine at any time. While lying in the MRI scanner, patients will be asked to perform tasks presented via a screen. These tasks will involve looking at pictures or words, and patients will be asked to make decisions about the pictures. The MRI scan will take no more than 2 hours. In regard to the computer-based tasks that participants will perform, the tasks are often games presented on a computer. Via computer, or on paper, there may be presentations of pictures that bring about an emotion.

There will be no direct treatment or therapeutic benefits to participation in this study. However, the knowledge gained may help people in the future.

DETAILED DESCRIPTION:
The Psychopathy Checklist-Revised (Hare, 1991) allows the identification of a relatively homogeneous population of individuals who present with marked emotional dysfunction (reduced empathy, guilt and attachment to others) as well as a notable propensity for goal-directed antisocial behavior. Identification of the neuro-biological underpinnings of their emotional dysfunction is of crucial importance as the level of emotion dysfunction is an important predictor of long term prognosis.

Currently, there are two main positions regarding the neural systems that are dysfunctional in individuals with psychopathy: First, that the pathology is associated with amygdala dysfunction; Secondly, that the pathology is associated with orbital frontal cortex dysfunction. A third, more recent position, stresses the interconnections between these two systems and the role that development may play in the disorder.

The current project will determine the performance of individuals with psychopathy and comparison individuals on measures which recruit the amygdala and orbital frontal cortex. In addition, a series of functional neuro-imaging studies will directly assess neural responses in these two systems in individuals with psychopathy. Finally, a structural imaging study will examine anatomical differences between the groups. The project should provide clear data that will constrain future theorizing on the pathology implicated in this disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Psychopathy:

     1. Comparison individuals: All individuals will score less than 20 on the PCL-R.
     2. Individuals with psychopathy: All individuals will score more than 30 on the PCL-R (participants scoring between 21-29 are excluded from study participation).
  2. Age: Participants will be males and females, 20-50 years of age.
  3. IQ: IQ, as measured by 4 subscales from the Wechsler Adult Intelligence Scale-Revised (WAIS-R), must be greater than 80.
  4. Medication status: No current use of any psychotropic medication or benzodiazepine.

EXCLUSION CRITERIA:

Because factors such as psychiatric disease, or CNS disease, can influence functional brain activity, these factors are exclusionary.

1. Psychiatric history: Participants will be assessed using DSM-IV criteria via standardized psychiatric interviews conducted by trained examiners (i.e., SCID).

   1. Comparison individuals: All participants will be free of any current or past psychiatric disorder. Participants will be excluded if they meet criteria for substance dependence but not if they meet criteria for substance abuse.
   2. Individuals with psychopathy: It is to be expected that the individuals with psychopathy will meet diagnostic criteria for Antisocial Personality Disorder and, in childhood, would have met criteria for Conduct Disorder, Oppositional Defiant Disorder and probably Attentional Deficit and Hyperactivity Disorder. Any other current or past psychiatric disorder will be exclusory. Participants will be excluded if they meet criteria for substance dependence but not if they meet criteria for substance abuse.
2. Severe acute and chronic medical illnesses. In short, any condition requiring the administration of systemic drugs will be exclusory.
3. CNS disease: history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), or other neurological disease, or history of head trauma (defined as loss of consciousness greater than 3 min).
4. Metal or electronic objects: Metal plates, certain types of dental braces, cardiac pacemakers, etc., that are sensitive to electromagnetic fields contraindicate MRI scans.
5. Claustrophobia: participants will be questioned about potential discomfort in being in an enclosed space, such as an MRI scanner.
6. There will be no exclusion criteria as regards type of crime. While there is some increase in risk to testers in having participants who have committed acts of violence, it is not extreme as long as the participants are appropriately treated. Indeed, in our previous work almost all of our participants (comparison individuals and individuals with psychopathy) were murderers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160
Dates: Start 2004-08-27; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Angrilli A, Mauri A, Palomba D, Flor H, Birbaumer N, Sartori G, di Paola F. Startle reflex and emotion modulation impairment after a right amygdala lesion. Brain. 1996 Dec;119 ( Pt 6):1991-2000. doi: 10.1093/brain/119.6.1991. PMID 9010003